CLINICAL TRIAL: NCT00238251
Title: Whole Brain Radiotherapy in Combination With Gefitinib (Iressa) or Temozolomide (Temodal) for Brain Metastases From Non-Small Lung Cancer (NSCLC) A Randomized Phase II Trial
Brief Title: Radiation Therapy Combined With Either Gefitinib or Temozolomide in Pats With NSCLC and Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 70/03; EU-20526
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; tumors metastatic to brain
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Gefitinib; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients undergo whole-brain radiotherapy (WBRT) once daily on days 1-5 and 8-12 and receive oral gefitinib once daily on days 1-28. Gefitinib treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: gefitinib; Radiation: radiation therapy
- Arm II (Active Comparator): Patients undergo WBRT as in arm I and receive oral temozolomide once daily on days 1-21. Temozolomide treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: temozolomide; Radiation: radiation therapy

INTERVENTIONS:
Drug: gefitinib — Once daily during days 1-28
  Arms: Arm I
Drug: temozolomide — Once daily on days 1-21
  Arms: Arm II
Radiation: radiation therapy — Whole brain radiotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with either gefitinib or temozolomide may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well giving radiation therapy together with either gefitinib or temozolomide works in treating patients with non-small cell lung cancer and brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of whole-brain radiotherapy combined with either gefitinib or temozolomide, in terms of overall survival, in patients with non-small cell lung cancer and brain metastases.

Secondary

* Compare the tolerability and toxicity of these regimens in these patients.
* Compare the time to neurological disease progression, time to extracranial disease progression, and time to overall disease progression, in patients treated with these regimens.
* Compare adverse events in patients treated with these regimens.
* Compare cognitive function and quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, parallel-group, multicenter study. Patients are stratified according to extracranial disease (yes vs no), number of brain metastases (1-3 vs ≥ 4), prior chemotherapy (yes vs no), WHO performance status (0-1 vs 2), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo whole-brain radiotherapy (WBRT) once daily on days 1-5 and 8-12 and receive oral gefitinib once daily on days 1-28. Gefitinib treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo WBRT as in arm I and receive oral temozolomide once daily on days 1-21. Temozolomide treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and on day 1 of courses 2, 3, and 5.

After completion of study therapy, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 30-86 patients (15-43 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer AND newly diagnosed brain metastases meeting 1 of the following criteria:

  * Multiple brain metastases
  * Single brain metastasis not amenable to potentially curative treatment
* No advanced extracranial disease severely compromising vital functions and performance

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin > 10 g/dL
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN (5 times ULN in the presence of documented bone metastases)
* No unstable or uncompensated hepatic disease that would preclude study participation

Renal

* Creatinine clearance ≥ 40 mL/min
* No unstable or uncompensated renal disease that would preclude study participation

Cardiovascular

* No myocardial infarction within the past 3 months
* No unstable or uncompensated cardiac disease that would preclude study participation

Pulmonary

* No clinically active interstitial lung disease

  * Patients with chronic stable radiographic changes who are asymptomatic eligible
* No other unstable or uncompensated respiratory disease that would preclude study participation

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* No nausea, vomiting, inability to swallow whole tablets/capsules, or malabsorption syndrome that would preclude oral medication ingestion or absorption
* No psychiatric disorder that would preclude giving informed consent or study compliance
* No active infection
* No uncontrolled diabetes mellitus
* No other medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior temozolomide

Endocrine therapy

* Concurrent corticosteroids allowed provided dose has been stable or decreasing for ≥ 4 days before study entry

Radiotherapy

* No prior brain irradiation

Surgery

* Not specified

Other

* No prior gefitinib or erlotinib
* More than 30 days since prior investigational clinical trial participation
* No other concurrent experimental drugs
* No other concurrent anticancer therapy
* No concurrent treatment with any of the following:

  * Phenytoin
  * Carbamazepine
  * Rifampin
  * Barbiturates
  * Hypericum perforatum (St. John's wort)
  * Other enzyme-inducing anti-epileptic drugs or tuberculostatic treatments
  * Any drug that contraindicates administration with study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2005-05; Primary Completion 2009-04 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | life-long

SECONDARY OUTCOMES:
Time to progression | 28 days
Time to neurological progression | 28 days
Time to extracranial disease progression | 28 days
Adverse events as measured at completion of study treatment | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Pesce, MD, Study Chair — Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni; Roger Stupp, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (3):
- Switzerland (3):
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Kantonsspital Graubuenden, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne

REFERENCES:
- [Result] Pesce GA, Klingbiel D, Ribi K, Zouhair A, von Moos R, Schlaeppi M, Caspar CB, Fischer N, Anchisi S, Peters S, Cathomas R, Bernhard J, Kotrubczik NM, D'Addario G, Pilop C, Weber DC, Bodis S, Pless M, Mayer M, Stupp R. Outcome, quality of life and cognitive function of patients with brain metastases from non-small cell lung cancer treated with whole brain radiotherapy combined with gefitinib or temozolomide. A randomised phase II trial of the Swiss Group for Clinical Cancer Research (SAKK 70/03). Eur J Cancer. 2012 Feb;48(3):377-84. doi: 10.1016/j.ejca.2011.10.016. Epub 2011 Nov 15. PMID 22093943